CLINICAL TRIAL: NCT05820607
Title: Clinical Characteristics, Lifestyle and Integrated Microbiome, Metabolome, Transcriptome, Genome Analysis in Autoimmune Gastritis
Brief Title: Clinical Characteristics, Lifestyle and Multi-omics Analysis in Autoimmune Gastritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Tong Ren Hospital (Other); Seventh Medical Center of PLA Army General Hospital (Other); Tianjin Medical University General Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Southern Medical University, China (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Jing-yuan Fang, MD, Ph. D, Director of Department of Gastroenterology of Renji Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: KY2022-134-B
Record Dates: First submitted 2023-03-23; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Autoimmune Gastritis
MeSH Terms: interventions — Microbiota; Metabolome; Transcriptome; Genome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood specimen, gastric mucosa biopsy tissue specimen and feces specimen
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type A atrophic gastritis: Gastroscopy and histopathology showed no significant atrophy of antrum mucosa, but significant atrophy of the body or fundus mucosa, accompanied by positive blood and/or gastric fluid anti-parietal cell antibodies and/or anti-internal factor antibodies.
  Interventions: Biological: Microbiome, metabolome, transcriptome, genome
- Type B atrophic gastritis: Gastroscopy and histopathological examination showed multifocal atrophy of gastric mucosa, mainly antrum involved.
  Interventions: Biological: Microbiome, metabolome, transcriptome, genome
- Chronic non-atrophic gastritis: Gastroscopy and histopathology showed chronic inflammation of gastric mucosa with infiltration of lymphocytes and plasma cells, and no intrinsic glandular reduction.
  Interventions: Biological: Microbiome, metabolome, transcriptome, genome

INTERVENTIONS:
Biological: Microbiome, metabolome, transcriptome, genome — Fecal genome, serum metabolome, leukocyte transcriptome, gastric mucosa genome

SUMMARY:
This research will be conducted nationwide in patients with autoimmune gastritis, focusing on their clinical characteristics, possible risk factors, and multi-omics analysis. Changes in gastrointestinal microbiota, host and microbial metabolism, gene transcription and biomarkers of autoimmune gastritis will be explored to provide evidence for further precise therapy of the disease.

DETAILED DESCRIPTION:
Autoimmune gastritis is a chronic progressive disease that may develop into gastric cancer. However, on account of its low morbidity, atypical clinical and endoscopic manifestation, demanding technique for detection of serological markers, the diagnosis and treatment of this disease remains challenging. Therefore, there's inadequate studies focusing on its pathogenesis, metabolism, gene transcription, microbiota etc. In recent years, multi-omics analysis provides clinicians with depth and breadth understandings of diseases. This research, as well, aims at enhancing clinicians' knowledge of autoimmune gastritis to reduce the occurrence of neuroendocrine tumors, gastric cancer, pernicious anemia and other complications.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35-75 years.
* Type A atrophic gastritis: Underwent gastroscopy in hospitals mentioned above. Gastroscopy and histopathology showed no significant atrophy of antrum mucosa, but significant atrophy of the body or fundus mucosa, accompanied by positive blood and/or gastric fluid anti-parietal cell antibodies and/or anti-internal factor antibodies. No obvious tumor, deep ulcer, severe bile reflux, severe erosion, or active bleeding. Type B atrophic gastritis: Underwent gastroscopy in hospitals mentioned above. Gastroscopy and histopathological examination showed multifocal atrophy of gastric mucosa, mainly antrum involved. No obvious tumor, ulcer, moderate to severe bile reflux, moderate to severe erosion, multiple polyps (≥2) , or active bleeding. Chronic non-atrophic gastritis: Underwent gastroscopy in hospitals mentioned above. Gastroscopy and histopathology showed chronic inflammation of gastric mucosa with infiltration of lymphocytes and plasma cells, and no intrinsic glandular reduction. No obvious tumor, ulcer, moderate to severe bile reflux, moderate to severe erosion, multiple polyps (≥2) , or active bleeding.
* Underwent colonoscopy within the past 5 years, and no obvious abnormalities such as inflammation, polyps, tumor, or ulcer were observed.
* Have the cognitive level to understand the questionnaire and cooperate voluntarily.

Exclusion Criteria:

* Aged <35 years or>75 years.
* Histopathology indicated dysplasia.
* Long-term use of PPIs or H2-blockers for more than 3 months in the past 1 year. With a history of Helicobacter pylori eradication within the past 2 months.
* Use of antibiotics, nonsteroidal anti-inflammatory drugs, probiotics, steroids, or immunosuppressants for more than 2 weeks within the past 2 months.
* Severe constipation or diarrhea within the past 3 months, or notable changes in bowel habits within the past 3 months.
* History of tumor, organ transplantation, or severe parasitic disease, other diseases of digestive system (such as inflammatory bowel disease, cirrhosis, pancreatitis, etc.), or serious infection.
* History of severe trauma, major operation, extensive burn, cerebral vascular accident, severe organ failure (cardiac, hepatic, renal insufficiency, etc.), shock or sepsis within the past 6 months.
* History of gastrointestinal surgery.
* History of gastrointestinal bleeding, ileus, perforation.
* Chronic metabolic, infectious, or endocrine diseases (such as hypertension, diabetes, hyperlipidemia, hyperuricemia, hyperpurine) that are not well controlled, whether or not treated with medications.
* Vegetarians or had significant changes in eating habits within the past 3 months.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese people
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-06-19 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Differences in microbiome | 1 year
  Differences in microbiome within or between groups will be explored by metagenomic sequencing and validated by molecular biology experiments
Differences in metabolome | 1 year
  Differences in microbiome within or between groups will be explored by mass spectrometry and validated by molecular biology experiments
Differences in transcriptome | 1 year
  Differences in microbiome within or between groups will be explored by transciptome sequencing and validated by molecular biology experiments
Differences in genome | 1 year
  Differences in microbiome within or between groups will be explored by 16s RNA sequencing and validated by molecular biology experiments

SECONDARY OUTCOMES:
Differences in clinical outcomes | 1 year
  Differences in clinical outcomes of Group 1, whether subjects have complications, such as folic acid or vitamin B12 deficiency (folic acid<3.1ug/L, vitamin B12<180pg/ml), anemia ( male Hb<130g/L, female Hb<115g/L), hyperplastic polyp, pseudopolyp, pyloric adenoma, type 1 neuroendocrine tumor or gastric cancer (pathologically confirmed), all these complications will be reported separately
Differences in lifestyle | 1 year
  Differences in lifestyle within or between groups acquired by food frequency questionnaire and analyzed by statistical approaches

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Fang, MD, Ph.D, Principal Investigator — Shanghai Institute of Digestive Disease
Locations (1):
- Shanghai Institute of Digestive Disease, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No